CLINICAL TRIAL: NCT04899349
Title: EPIK-B4: A Phase II, Multicenter, Randomized, Open-label, Active-controlled Study to Assess the Safety and Efficacy of Dapagliflozin + Metformin XR Versus Metformin XR During Treatment With Alpelisib (BYL719) in Combination With Fulvestrant in Participants With HR+, HER2-, Advanced Breast Cancer With a PIK3CA Mutation Following Progression on/After Endocrine-based Therapy
Brief Title: Study of Safety and Efficacy of Dapagliflozin + Metformin XR Versus Metformin XR in Participants With HR+, HER2-, Advanced Breast Cancer While on Treatment With Alpelisib and Fulvestrant
Acronym: EPIK-B4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was early terminated due to slow recruitment and emerging data showing that prophylactic use of metformin may prevent or reduce the incidence of all-grades alpelisib-related hyperglycemia. The decision was not driven by safety concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CBYL719C2202
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Alpelisib; Fulvestrant; Metformin XR; Dapagliflozin + metformin XR; Advanced breast cancer; Phase II; HR+; HER2-; PIK3CA; Hyperglycemia
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies; Hyperglycemia | interventions — Alpelisib; Fulvestrant; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR (Experimental): Alpelisib 300mg administered orally once daily starting at Cycle 1 Day 8 in combination with fulvestrant 500mg intramuscular at Cycle 1 Day 1 and 15 and then at Day 1 of each subsequent cycle. Participants also received a combination treatment of dapagliflozin+metformin XR (as a single tablet or as two separate tablets, at the discretion of the investigator) at a starting dose of 5 mg dapagliflozin + 500 mg metformin XR orally once daily which could be titrated to a maximum dose of 10 mg dapagliflozin + 2000 mg metformin XR once daily.
  Interventions: Drug: Alpelisib; Drug: Fulvestrant; Drug: Metformin XR; Drug: Dapagliflozin + metformin XR; Drug: Dapagliflozin
- Alpelisib + Fulvestrant + Metformin XR (Active Comparator): Alpelisib 300mg administered orally once daily starting at cycle 1 Day 8 in combination with fulvestrant 500mg intramuscular at Cycle 1 Day 1 and 15 and then at Day 1 of each subsequent cycle. Participants also received metformin XR 500mg orally once daily which could be titrated to a maximum dose of 2000 mg once daily.
  Interventions: Drug: Alpelisib; Drug: Fulvestrant; Drug: Metformin XR

INTERVENTIONS:
Drug: Alpelisib — Alpelisib (tablets) administered at 300mg orally once daily on a continuous dosing schedule starting on Cycle 1 Day 8 in a 28 days cycle.
Drug: Fulvestrant — Fulvestrant (prefilled syringe) 500mg administered intramuscularly at Cycle 1 Day 1 and 15 after randomization and then at Day 1 of each subsequent cycle during the randomized treatment phase.
Drug: Metformin XR — Metformin XR (tablets) administered at a starting dose of 500mg orally once daily on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28 days cycle. Dose titration from 500 mg once a day to 2000 mg once a day.
Drug: Dapagliflozin + metformin XR — Dapagliflozin + metformin XR administered as a single tablet combination at a starting dose of 5 mg dapagliflozin + 500 mg metformin XR orally once daily on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28 days cycle. Dose titration from 5 mg dapagliflozin + 500 mg metformin XR orally once daily to 10 mg dapagliflozin + 2000 mg metformin XR once daily
  Arms: Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR
Drug: Dapagliflozin — Dapagliflozin (tablet) at a starting dose of 5mg orally once daily on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28 days cycle. Dose titration from 5 mg to 10 mg once daily
  Arms: Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR

SUMMARY:
This study was designed to assess the safety and efficacy of the combination of dapagliflozin plus metformin extended release (XR) compared with metformin XR during treatment with alpelisib plus fulvestrant in participants with Hormone Receptor (HR)-positive, Human Epidermal growth factor Receptor-2 (HER2)-negative advanced breast cancer with a Phosphoinositide-3-Kinase Catalytic subunit Alpha (PIK3CA) mutation following progression on or after endocrine-based therapy.

DETAILED DESCRIPTION:
This was a multicenter, randomized, open-label, active-controlled trial, stratified by diabetic status at baseline (i.e., normal vs prediabetic/diabetic based on fasting plasma glucose (FPG) and/or Hemoglobin A1c (HbA1c) laboratory values). The study included only participants with at least one baseline risk factor for the development of severe hyperglycemia which were diabetes (FPG ≥ 126 milligram (mg)/deciliter (dL) or ≥ 7.0 millimole (mmol)/liter (L) and/or HbA1c ≥ 6.5%), prediabetes (FPG ≥ 100 mg/dL to < 126 mg/dL or 5.6 to < 7.0 mmol/L and/or HbA1c 5.7 to < 6.5%), obesity (body mass index [BMI] ≥ 30) and age (≥ 75 years).

The planned duration of treatment with alpelisib and fulvestrant was 12 cycles (28 days in each cycle) or until disease progression, unacceptable toxicity, or discontinuation from study treatment for any other reason, whichever came first.

Approximately 66 participants in each treatment arm were planned to be randomized to receive the combination of alpelisib and fulvestrant with either dapagliflozin plus metformin extended release (XR) or metformin XR alone. As a result of the early termination of the study due to emerging data demonstrating the impact of prophylactic metformin and slow recruitment, only 2 participants were enrolled in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant had a histologically and/or cytologically confirmed diagnosis of estrogen receptor positive (ER+) and/or progesterone receptor positive (PgR+) breast cancer by a local laboratory.
* Participant had a PIK3CA mutation(s) present in the tumor prior to enrollment.
* Participant had prior treatment with an endocrine-based treatment (e.g. letrozole, anastrozole, exemestane, fulvestrant, or oral SERD) and may have fallen into one of the following categories:

  1. Relapsed with documented evidence of progression while on (neo) adjuvant endocrine-based therapy or within 12 months from completion of (neo) adjuvant endocrine-based therapy with no treatment for metastatic disease.
  2. Relapsed with documented evidence of progression more than 12 months from completion of (neo) adjuvant endocrine-based therapy and then subsequently progressed with documented evidence of progression while on or after only one line of endocrine-based therapy for metastatic disease.
  3. Newly diagnosed advanced breast cancer, then relapsed with documented evidence of progression while on or after only one line of endocrine-based therapy.

Note: Participants with newly diagnosed endocrine-based treatment naïve advanced breast cancer were NOT included in the study.

* Participants might or might not have received prior CDK4/6i therapy. If prior CDK4/6i therapy was administered, it may have been in the adjuvant or metastatic setting.
* If female, the participant was postmenopausal.
* Participant had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participant had adequate bone marrow and organ function.

Key Exclusion Criteria:

* Participant relapsed with documented evidence of progression more than 12 months from completion of (neo) adjuvant endocrine therapy with no treatment for metastatic disease.
* Participant had more than 1 line of prior treatment in the metastatic setting.
* Participant had received prior treatment with chemotherapy (except for neoadjuvant/adjuvant chemotherapy), any PI3K, Mammalian Target of Rapamycin (mTOR) or Protein Kinase B (Akt) inhibitor.
* Participant had inflammatory breast cancer at screening.
* Participants with an established diagnosis of diabetes mellitus type I or participants with type II diabetes mellitus requiring antihyperglycemic therapy.
* Participant had a history of acute pancreatitis within 1 year of screening or a past medical history of chronic pancreatitis.
* Participant had currently documented pneumonitis/interstitial lung disease.
* Participant had a history of severe cutaneous reaction, such as Steven-Johnson Syndrome (SJS), erythema multiforme (EM), Toxic Epidermal Necrolysis (TEN) or Drug Reaction with Eosinophilia and Systemic Syndrome (DRESS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Washington Uni School of Med Siteman Cancer Center, St Louis, Missouri, United States
- Novartis Investigative Site, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 sites in 2 countries enrolled participants
Pre-assignment Details: Screening assessments were conducted up to 21 days prior to the randomization. The trial was early terminated and no patients were randomized to the Alpelisib + Fulvestrant + Metformin XR arm.
Period: Overall Study
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Study terminated by Sponsor | 2 | 0

BASELINE CHARACTERISTICS:
Population: The trial was early terminated and no participants were randomized to the Alpelisib+Fulvestrant+Metformin XR arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70 (4.24) |  | 70 (4.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hyperglycemia Grade ≥ 3 Over the First Eight Weeks of Alpelisib Plus Fulvestrant Treatment
Description: Number of participants with severe hyperglycemia over the first eight weeks of alpelisib plus fulvestrant treatment. Severe hyperglycemia (Grade ≥ 3) is defined as any glucose laboratory values > 250 milligram (mg)/ deciliter (dL) (> 13.9 millimole (mmol)/ liter (L))
Time Frame: From Cycle 1 Day 8 to Cycle 3 Day 8 (first eight weeks of treatment with alpelisib). Cycle = 28 days.
Population: All participants who received at least one dose of study treatment (i.e. at least one dose of any component of alpelisib, fulvestrant, dapagliflozin + metformin XR, metformin XR).
  The trial was early terminated and no participants were randomized to the Alpelisib + Fulvestrant + Metformin XR arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR
Number analyzed (Participants) | 2 | 0
Participants | 1 |

2. Secondary Outcome: Progression-free Survival (PFS) Based on Local Investigator Assessment
Description: PFS was defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. PFS was assessed via a local investigator assessment according to RECIST 1.1. If a subject did not have an event, PFS was censored at the date of last adequate tumor assessment.
  The PFS distribution was using the Kaplan-Meier method, and the Kaplan-Meier median and 95% confidence intervals of the medians was presented.
Time Frame: From the date of randomization to the date of the first documented progression or death due to any cause, whichever comes first, assessed up to a maximum duration of 7.4 months
Population: All participants to whom study treatment was assigned by randomization. The trial was early terminated and no participants were randomized to the Alpelisib + Fulvestrant + Metformin XR arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR
Number analyzed (Participants) | 2 | 0
Months | NA [NA to NA] — NA. Not estimable as none of the participants had an event |

3. Secondary Outcome: Overall Response Rate (ORR) With Confirmed Response Based on Local Investigator Assessment as Per RECIST 1.1.
Description: ORR with confirmed response was defined as the percentage of participants with best overall response of confirmed complete response (CR) or confirmed partial response (PR) based on local investigator's assessment according to RECIST 1.1.
  CR: Disappearance of all non-nodal target lesions and all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions and all lymph nodes assigned as non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 7.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR
Number analyzed (Participants) | 2 | 0
Participants | 1 |

4. Secondary Outcome: Clinical Benefit Rate (CBR) With Confirmed Response Based on Local Investigator Assessment as Per RECIST 1.1
Description: Clinical benefit rate with confirmed response was defined as the percentage of participants with a best overall response of confirmed CR or confirmed PR or stable disease (SD) or Non-CR/Non-progressive disease (PD) lasting more than 24 weeks based on local investigator assessment as per RECIST 1.1.
  CR: Disappearance of all non-nodal target lesions and all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions and all lymph nodes assigned as non-target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to 7.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR
Number analyzed (Participants) | 2 | 0
Participants | 1 |

5. Secondary Outcome: Number of Participants With Dose Modifications
Description: Number of participants with dose interruptions and dose reductions
Time Frame: From first dose of study medication up to 30 days after last dose of study medication, assessed up to 7.4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR
Number analyzed (Participants) | 2 | 0
Participants
  Dose interruptions | 1 | 0
  Dose reductions | 2 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study medication up to 30 days after last dose of study medication, assessed up to 7.4 months
Description: All participants who received at least one dose of study treatment (i.e. at least one dose of any component of alpelisib, fulvestrant, dapagliflozin + metformin XR, metformin XR).
  The trial was early terminated and no participants were randomized to the Alpelisib + Fulvestrant + Metformin XR arm.
Arm/Group | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR | Alpelisib + Fulvestrant + Metformin XR
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alpelisib + Fulvestrant + Dapagliflozin + Metformin XR (N=2) | Alpelisib + Fulvestrant + Metformin XR (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | NA
Constipation (Gastrointestinal disorders) | 2 | NA
Diarrhoea (Gastrointestinal disorders) | 1 | NA
Dry mouth (Gastrointestinal disorders) | 1 | NA
Nausea (Gastrointestinal disorders) | 2 | NA
Stomatitis (Gastrointestinal disorders) | 1 | NA
Vomiting (Gastrointestinal disorders) | 1 | NA
Fatigue (General disorders) | 2 | NA
Peripheral swelling (General disorders) | 1 | NA
Hypersensitivity (Immune system disorders) | 1 | NA
Blood cholesterol increased (Investigations) | 1 | NA
Blood creatinine increased (Investigations) | 1 | NA
Weight decreased (Investigations) | 1 | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | NA
Taste disorder (Nervous system disorders) | 1 | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | NA
Hot flush (Vascular disorders) | 1 | NA
Hypertension (Vascular disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT04899349/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT04899349/SAP_001.pdf